CLINICAL TRIAL: NCT07333144
Title: Management of Gastrointestinal Bleeding Under Direct Oral Anticoagulants: Analysis of Reversal Practices Using Prothrombin Complex at the Strasbourg University Hospitals
Brief Title: Management of Gastrointestinal Bleeding Under Direct Oral Anticoagulants
Acronym: HEMOD-AOD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9612
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Bleeding
Keywords: Gastrointestinal bleeding; Hepatogastroenterology; Direct oral anticoagulants
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal bleeding (GIB) is a common emergency in hepatology and gastroenterology, with an overall mortality rate ranging from 5% to 10% depending on the study. GIB is classified into two categories: upper GIB (80% of cases) and lower GIB (20% of cases). There are many risk factors for GIB, including anticoagulants. In cases of GD under anticoagulants, there are specific management recommendations. In particular, in cases of severe bleeding under direct oral anticoagulants (DOACs), it is recommended to stop treatment and correct coagulation parameters according to the severity of the bleeding and the associated thrombotic risk. Various treatments can be used for this purpose, including specific antidotes, fresh frozen plasma, and prothrombin complex concentrate (PCC). However, the role of PCC in this indication is uncertain, as is the efficacy and safety data for this drug, due to significant methodological limitations in the few studies conducted on the subject.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Male or female
* Patient admitted to the emergency department for gastrointestinal bleeding (hematemesis, melena, rectal bleeding, or hematochezia)
* Taking a direct oral anticoagulant (dabigatran, apixaban, or rivaroxaban)

Exclusion Criteria:

* Subject who has expressed their objection to the reuse of their data for scientific research purposes.
* Subject under guardianship, curatorship, or legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years) admitted to the emergency department for gastrointestinal bleeding (hematemesis, melena, rectal bleeding, or hematochezia) and aking a direct oral anticoagulant (dabigatran, apixaban, or rivaroxaban)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients on direct oral anticoagulants admitted to the emergency department of Strasbourg University Hospital | 48 hours following patient admission
  Proportion of patients on direct oral anticoagulants admitted to the emergency department of Strasbourg University Hospital for gastrointestinal bleeding who received prothrombin complex concentrate within the first 48 hours of admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Urgences Adultes - CHU de Strasbourg - France, Strasbourg, France